CLINICAL TRIAL: NCT04634929
Title: Changes in Endocrinological and Central Neuronal Satiety Regulation Following Bariatric Surgery
Brief Title: Endocrinological and Neuronal Aspects of Bariatric Surgery
Acronym: BACEN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Heidelberg Medical Center (Other)
Responsible Party: Principal Investigator, Joe Simon, Principal Investigator, University of Heidelberg Medical Center
Other Study IDs: S-656/2019
Record Dates: First submitted 2020-11-03; First posted 2020-11-18 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Bariatric Surgery; Obesity
Keywords: fMRI; hormonal satiety signaling; hypothalamus; weight loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- bariatric surgery participants: participants with obesity planning to undergo bariatric surgery
  Interventions: Procedure: bariatric surgery
- conservative diet participants: participants with obesity planning to controlled conservative behavioral weight loss program
  Interventions: Dietary Supplement: conservative diet

INTERVENTIONS:
Procedure: bariatric surgery — bariatric surgery
  Groups: bariatric surgery participants
Dietary Supplement: conservative diet — conservative diet
  Groups: conservative diet participants

SUMMARY:
The overall aim of the proposed project is to investigate the contribution of changes in neuronal food processing, hypothalamic reactivity and hormonal factors to weight loss after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* planning to undergo bariatric surgery
* planning to take part in a conservative diet

Exclusion Criteria:

* inability to undergo fMRI
* psychiatric disorders
* metabolic disorders

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: healthy participants with obesity
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Change in Functional magnetic resonance imaging following intravenous glucose infusion. | 2 weeks before surgery or start of dietary intervention and 2 weeks after surgery or start of dietary intervention.
  Change in responsivity of the hypothalamus (extracted as percent signal change) as the core region of homeostatic control will be assessed after an intravenous glucose infusion (by calculating the area under the curve of hypothalamic responsivity) before and after bariatric surgery or dietary intervention.
Experimental functional magnetic resonance imaging task (gustatory stimulation). | 2 weeks before surgery or start of dietary intervention and 2 weeks after surgery or start of dietary intervention.
  Neuronal gustatory processing of food stimuli will be assessed (ingestion of sweet liquids using a gustometer) using a general linear model (comparing brain activation during ingestion of sweet liquids with brain activation during the ingestion of water) and within as well as between groups analyses. Changes in neural gustatory processing of food stimuli will be assessed before and after bariatric surgery or dietary intervention.
Assessment of glucose-induced changes in peripheral ghrelin using blood samples. | 15 minutes before and 15 minutes after functional magnetic resonance imaging
  Blood is collected to measure the concentration of peripheral ghrelin as an indicator of hormonal satiety signaling. Blood samples are collected at the beginning and end of each experimental session to assess the influence of intravenuous infusion of glucose on ghrelin signaling. Blood samples will be analysed using using commercially available kits (enzyme-linked immunosorbent assay).

OTHER OUTCOMES:
Weight change | 12 months
  Change in weight following bariatric surgery or dietary intervention

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Billeter, PD, MD, Principal Investigator — Department of General, Visceral, and Transplantation Surgery, University of Heidelberg
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No
upon reasonable request